CLINICAL TRIAL: NCT02570204
Title: Self-Assessment of Medical Abortion Outcome Using Serial Multi-level Pregnancy Tests
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1033
Record Dates: First submitted 2015-10-05; First posted 2015-10-07 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Medical Abortion
MeSH Terms: interventions — Diagnostic Self Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Self-assessment of abortion outcome (Experimental): Patients enrolled in the study will self-assess the outcomes of their medical abortion with the aid of a multi-level pregnancy test (MLPT) which they will perform at home.
  Interventions: Behavioral: Self-assessment

INTERVENTIONS:
Behavioral: Self-assessment — Patients enrolled into the study will do a multi-level pregnancy test (MLPT) at enrollment, and will receive one MLPT to do at home one week after taking mifepristone and misoprostol. They will be instructed to call the study site if the at-home MLPT result do not decline, or if they experience any abortion complications.

SUMMARY:
This study aims to investigate the effectiveness and acceptability of the multi-level pregnancy test for self-assessment of abortion outcomes, without a routine provider contact.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age of less than or equal to 63 days
* Determined by the site investigator or designee to be fully eligible for medical abortion with mifepristone followed by misoprostol according to the site's standard criteria
* Willing to use the MLPT at home
* 11-56 years old
* Willing and able to comply with study procedures
* In the judgement of the site investigator, she is capable of giving informed consent and she has signed the study informed consent or assent form

Exclusion Criteria:

-

Ages: 11 Years to 56 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 343 (Actual)
Dates: Start 2015-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who fail to contact the clinic when indicated within two weeks after taking the mifepristone | One month

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Raymond, MD, MPH, Study Director — Gynuity Health Projects
Locations (3):
- United States (3):
  - Presidential Women's Center, West Palm Beach, Florida
  - Carafem, Chevy Chase, Maryland
  - Philadelphia Women's Center, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Raymond EG, Tan YL, Grant M, Benavides E, Reis M, Sacks DN, Hannum C, Frapp S, Weaver MA. Self-assessment of medical abortion outcome using symptoms and home pregnancy testing. Contraception. 2018 Apr;97(4):324-328. doi: 10.1016/j.contraception.2017.12.004. Epub 2017 Dec 11. PMID 29242085